CLINICAL TRIAL: NCT03870087
Title: A Post-Market Study in Japan for the Evaluation of the CorPath® GRX System Effectiveness in Percutaneous Coronary Interventions
Brief Title: PRECISION GRX Post-Market Study - Japan
Status: Completed | Type: Observational
Sponsor: Corindus Inc. (Industry)
Collaborators: Japan Medicalnext, Co (Unknown)
Responsible Party: Sponsor
Other Study IDs: 104-08185
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Robotic PCI: All subjects treated with CorPath GRX during the PCI procedure.
  Interventions: Device: Robotic-assisted PCI

INTERVENTIONS:
Device: Robotic-assisted PCI — The CorPath GRX is intended for use in the remote delivery and manipulation of guidewires and rapid exchange balloon/stent catheters, and remote manipulation of guide catheters during percutaneous coronary intervention (PCI) procedures.

SUMMARY:
To collect data on the routine patterns of use, safety and effectiveness, including the clinical and technical performance of the CorPath GRX System, in the delivery and manipulation of coronary guidewires and stent/balloon catheters, and manipulation of guide catheters during PCI procedures in the first 231 patients treated with the CorPath device in Japan.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multi-center patient registry in Japan of the CorPath GRX System to examine its performance during PCI procedures and patient outcomes through 72 hours post-procedure or hospital discharge, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years;
2. Patients with coronary artery disease with clinical indication for PCI;
3. Patient deemed appropriate for robotic-assisted PCI; and
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, unless the EC has waived informed consent.

Exclusion Criteria:

1. Failure/inability/unwillingness to provide informed consent, unless the EC has waived informed consent; or
2. The Investigator determines that the patient or the coronary anatomy is not suitable for robotic-assisted PCI.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease and with a clinical indication for PCI.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Residual stenosis in the lesion(s) treated | Through end of subject's participation in the study, an average of up to 3 days.
  Less than 30% residual stenosis (visual estimate) post PCI in the lesion(s) treated with the CorPath GRX System, without in-hospital major adverse cardiac events (MACE) as assessed by the Angiographic Core Laboratory (ACL).
Technical Success | During procedure
  Defined as successful completion of the robotic-assisted PCI absent unplanned conversion to manual for guidewire or balloon/stent catheter inability to navigate vessel anatomy or poor guide catheter support.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | Through end of subject's participation in the study, an average of up to 3 days.
  MACE that occurs within 72 hours of the procedure or prior to hospital discharge, whichever occurs first, in a subject treated with the CorPath GRX System.
Overall Procedure Time | During procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
PCI Procedure Time | During procedure
  Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
IVUS/OCT/IVUS-OCT Time (if used) | During procedure
  Defined as the total time measured from insertion of the imaging catheter [Intravascular Ultrasound (IVUS), Optical Coherence Tomography (OCT) or integrated IVUS-OCT (IVUS-OCT)] until the removal of the imaging catheter.
Fluoroscopy Time | During procedure
  Total fluoroscopy utilized during the procedure as recorded by an Imaging System.
Patient Radiation Exposure | During procedure
  DAP (dose-area-product) and cumulative dose/air kerma as recorded during the procedure.
Operator Radiation Exposure | During procedure
  Cumulative dose the physician receives as recorded from electronic pocket dosemeter during procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, MD, Principal Investigator — Division of Cardiovascular Medicine, Professor Toho University Ohashi Medical Center
Locations (8):
- Japan (8):
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Nayoro City General Hospital, Nayoro, Hokkaido
  - Iwate University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Toho University Ohashi Medical Center, Tokyo, Ohashi Meguro-ku
  - Dokkyo Medical University Hospital, Mibu, Tochigi
  - Keio University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No